CLINICAL TRIAL: NCT04357652
Title: Contraception and Cervical and Breast Cancer Screening in Obese Versus Non-obese Women Aged 25 to 74 Years Old
Brief Title: Contraception and Cervical and Breast Cancer Screening in Obese Versus Non-obese Women
Acronym: DEPISGYN
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0130
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Obesity
Keywords: breast cancer; cervical cancer; contraception; screening
MeSH Terms: conditions — Obesity; Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
.Brief Summary:* Obesity is a major public health problem in France. Indeed, 17% of the French population is obese (BMI greater than or equal to 30 kg/m²) while almost half of the adult population is overweight (BMI greater than or equal to 25 kg/m²).

There is an increased risk of gynecological cancer in obese women but screening is less often performed :

In women, obesity is a risk factor for the occurrence of certain cancers such as uterine cancer, epithelial ovarian cancer and breast cancer, particularly post-menopausal. In addition, an increase in BMI from the first stage of obesity is associated with larger breast tumors with more frequent lymph node involvement, indicating more invasive cancers. Recent studies have shown an increase in breast cancer mortality for women with grade 2 and 3 obesity compared to women of so-called normal weight. Mortality from invasive breast cancer is higher from the obesity stage onwards.

The current recommendations of the High Authority for Health recommend breast cancer screening by mammography and clinical examination every two years in all women aged 50 to 74, excluding women at high risk and requiring specialist follow-up. Organized screening for cervical cancer has recently been modified. From 25 to 30 years of age the modalities remain the same and consist of two cytological examinations one year apart and then every 3 years if the latest results are normal. From the age of 30 and up to the age of 65, it is now recommended that an HPV test be performed as a first-line test, 3 years after the last normal cytological examination and then every 5 years if the last test was negative.

Studies dating back quite some time had shown an under-screening of cancers in obese women, in terms of carrying out mammography and cervical smears compared to women of normal weight. More recent data on access to gynecological cancer screening for obese women are heterogeneous, but there still seems to be less access to these examinations, whether for mammography or cervical smears. For example, a large American cohort study observed poorer detection of pre-cancerous lesions by smear with increasing BMI. Obese women had the lowest cumulative risk of pre-cancerous lesions at five years (followed by overweight women), but the highest rate of cancer at five years, associated with higher mortality.

A neglected contraception in obese women?

Data in the literature show that rates of unintended and unplanned pregnancies are higher in obese women (mainly those with grade 3 obesity) than in normal-weight women. This is associated with a lower use of contraception which is certainly poly-factorial: contraception not necessary due to a decrease in fertility linked to obesity, increased risks linked to contraception in obese women... However, most current contraceptive methods have shown similar efficacy in obese and non-obese women.

This context suggests that there is still a marked difference in the gynecological management of obese women. The role of the general practitioner seems essential in this follow-up by facilitating the use of screening tests and by improving the information of this population with regard to contraception in particular.

The objective of this study is to compare the gynecological follow-up of obese and non-obese women in a sample of women in Occitania, in terms of screening for breast and cervical cancer, as well as in terms of access to a method of contraception in general practice.

ELIGIBILITY:
Inclusion criteria:

* women from 25 to 74 years old
* BMI ≥ 18,5
* agree to participate in the study when they consult their endocrinologist or general practitioner.

Exclusion criteria:

* Subject opposition
* Subject in guardianship or trusteeship
* Women < 25 years of age and > 74 years of age
* Women with a BMI < 18.5 kg/m2
* Women with a history of breast or cervical cancer or hysterectomy.

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women between 25 and 74 years old, who have a consultation at the CHU of Montpellier in endocrinology and/or in metabolic surgery and/or in a general practice in Occitania for a period of 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of mammography screening | 1 day
  Rate of mammography screening in the previous two years among 50-74 year olds
Rate of screening by Pap smear or HPV test | 1 day
  Rate of screening by Pap smear or HPV test in the previous three years for 25-65 year olds.

SECONDARY OUTCOMES:
Rate of contraceptive prescriptions | 1 day
  Rate of contraceptive prescriptions among women aged 25 to 50.

CONTACTS AND LOCATIONS:
Overall Officials: Ariane SULTAN, PR, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC